CLINICAL TRIAL: NCT04262908
Title: Socio-professional Categories and Return to Work After Hip or Knee Replacement Surgery
Acronym: ARRET-Pro
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Responsible Party: Principal Investigator, Wilfrid GRAFF, Orthopedic surgeon, Groupe Hospitalier Diaconesses Croix Saint-Simon
Other Study IDs: ID RCB : 2019-A00046-51
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Hip Arthropathy Associated With Other Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients implanted with hip or knee prostheses: Patients who had hip or knee arthroplasty will be followed and asked at 3-months visit if they resumed their job or not. In both cases, further informations will be gathered
  Interventions: Other: Telephone call

INTERVENTIONS:
Other: Telephone call — Patients who did not return to work after the SL prescribed initially and had an extension of the SL will be called at 4 months postoperatively to collect infomation

SUMMARY:
A significant proportion of patients (15 to 45%) who have benefited from a total hip or knee replacement surgery (THKA), are put on sick leave (SL). This SL allows these patients who had a professional activity at the time of the intervention (age <65 years) to enhance the healing, improve the quality of life and ensure a functional return to work. The number of patients returning to work and the time taken to return to work after the intervention are d depending on the intervention (hip or knee) and are linked to socio-demographic factors, to the patient's general condition (comorbidity, presence of other arthritis joints…) and the type of professional activity.

Studies evaluating the impact of the type of professional activity on the return to work after THKA are nonexistent in France, rare in the literature, mostly retrospective and methodologically weak. In addition, the individual and socioeconomic impact of the cessation of work after an THKA, the absence of national data assessing the predictive nature of socio-professional categories on the return to work using a multivariate analysis motivated us to set up this study.

DETAILED DESCRIPTION:
The data usually collected in the medical file will be collected as part of the preoperative and 3 months postoperative study. As part of this study, a phone call will be made to contact patients who have had a prolonged SL

The data collected are as follows:

During hospitalization Socio-demographic data: sex, age, title of the profession, the joint concerned, family situation, place of life, postoperative availability of a caregiver or home help if necessary.

Clinical data: Comorbidities, weight, height, date of the arthroplasty, per and or postoperative complications of the arthroplasty, date of prescribed work stoppage

3 months postoperative: medical consultation Date of the 3-month consultation, date and method of resumption of work, if applicable, otherwise the duration of the extension of the duration of the SL, the doctor prescribing the extension and the causal link of this extension to the arthroplasty

4 months postoperative: telephone call This phone call will relate to patients whose work stoppage has been extended. Will be collected, the date and the mode of resumption of work, if not the cause of not resumed.

For patients whose prolongation of SL has been prescribed by the attending physician, the doctor of the rehabilitation center (knee prostheses) or by the occupational physician, the latter will be contacted by telephone to collect the reason for prolongation of the TA.

ELIGIBILITY:
Inclusion Criteria:

* Information of the patient and obtaining his non-opposition
* Men and women aged ≥ 18 and ≤ 65 and in full-time or part-time paid or voluntary professional activity before the intervention or before the work stoppage justified by the planned arthroplasty
* Patients consulting our orthopedic surgery department for the first implantation of a hip or knee prosthesis following arthritis

Exclusion Criteria:

* The patient expresses his opposition to the use of his personal data
* Patient> 65 years' old
* Arthroplasty on septic arthritis
* Presence of another hip or knee prosthesis already implanted
* Radiological stage 4 of osteoarthritis of the knee or hip not operated
* ASA > 3
* Proven depression or patient under antidepressant treatment
* Bipolarity, psychosis and neuroleptic treatment
* Retired patient
* Patient on sick leave ≥ 1 month before the intervention

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients consulting our orthopedic surgery department for a first total hip or knee arthroplasty who meet the study selection criteria The total number of inclusions is estimated at 300 patients.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Identification of socio-professional categories according to the PCS-ESE 2017 classification which would influence the return to work. | Through study completion, an average of 21 months
  To respond to the main objective of the study, investigator will collect
  ○ socio-demographic data during the anamnesis (sex, profession, joint concerned (hip, knee), family situation, place of life, presence of caregiver, co-morbidities, presence of other joint prostheses.
  * Clinical data (weight, height, musculoskeletal examination for other arthritis joints)
  * Data during hospitalization (date of surgery, intraoperative or postoperative complications (dislocation of prosthesis, bone or prosthesis stem fracture, hematoma, prosthesis infection)
  * Data concerning the work stoppage at 3 months during the usual follow-up consultation and by telephone as part of the study intervention about patients who have had a work stoppage extension (date of stoppage of work, date of resumption of work and mode of resumption, duration of extension of the SL, etc)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfrid GRAFF, MD, Principal Investigator — Groupe Hospitalier Diaconesses Croix Saint-Simon
Locations (1):
- Groupe Hospitalier Diaconesses Croix saint Simon, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tilbury C, Schaasberg W, Plevier JW, Fiocco M, Nelissen RG, Vliet Vlieland TP. Return to work after total hip and knee arthroplasty: a systematic review. Rheumatology (Oxford). 2014 Mar;53(3):512-25. doi: 10.1093/rheumatology/ket389. Epub 2013 Nov 23. PMID 24273048
- [Background] Tilbury C, Leichtenberg CS, Tordoir RL, Holtslag MJ, Verdegaal SH, Kroon HM, Nelissen RG, Vliet Vlieland TP. Return to work after total hip and knee arthroplasty: results from a clinical study. Rheumatol Int. 2015 Dec;35(12):2059-67. doi: 10.1007/s00296-015-3311-4. Epub 2015 Jun 29. PMID 26119221